CLINICAL TRIAL: NCT02492022
Title: A Double-blind Randomized Placebo-controlled Trial Assessing the Effectiveness of Two Probiotic Products During Nicotine Replacement Therapy for Managing Withdrawal Symptoms Associated With Smoking Cessation
Brief Title: Efficacy of 2 Probiotics During Nicotine Replacement Therapy on Withdrawal Symptoms Associated With Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Collaborators: MedQualis (Industry); Q & T Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Smoking Cessation
Record Dates: First submitted 2015-06-17; First posted 2015-07-08 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Probiotic L008-1 (Experimental): Encapsuled combinaison of 2 probiotics
  Interventions: Dietary Supplement: Probiotic L008-1
- Probiotic L008-2 (Experimental): Encapsuled combinaison of 2 probiotics
  Interventions: Dietary Supplement: Probiotic L008-2
- Placebo (Placebo Comparator): Encapsuled non active ingredients
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic L008-1 — Dosing regimen of 2 capsules daily, once per day, for 14 weeks
  Arms: Probiotic L008-1
Dietary Supplement: Probiotic L008-2 — Dosing regimen of 2 capsules daily, once per day, for 14 weeks
  Arms: Probiotic L008-2
Other: Placebo — Dosing regimen of 2 capsules daily, once per day, for 14 weeks
  Arms: Placebo

SUMMARY:
Quitting smoking is a big decision, a decision to achieve better health. Trying to quit smoking can be stressful. The prospect of dealing with withdrawal symptoms, fear or failure to change the routine, can also be sources of stress.

Withdrawal from nicotine is characterized by symptoms that include anxiety, irritability, hunger and cravings for more tobacco. Nicotine creates a dependency so that the body develops a need for a certain level of nicotine at all times. Unless that level is maintained symptoms of withdrawal appear.

For tobacco users trying to quit, symptoms of withdrawal from nicotine are unpleasant and stressful, but they are temporary.

Research has demonstrated the relative effectiveness of pharmacotherapy treatments in smoking cessation but no studies have examined the effects of the probiotics on the withdrawal symptoms associated with the tobacco cessation during nicotine replacement therapy (NRT).

The purpose of this study is to assess the effectiveness of two probiotic products during NRT for managing withdrawal symptoms associated with smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Moderate or heavy smokers as defined by:

a score at the Fargerström Test for Nicotine Dependence ≥ 5, and who smoke more than 10 cigarettes per day.

* Participants willing to stop smoking, corresponding to a score of 6 or 7 to the Motivation To Stop Scale. The MTSS is a one-item questionnaire with 7 possible choices, from 1 (lowest level of motivation to stop smoking) to level 7 (highest level of motivation to stop smoking).
* Participants need to be able to understand and consent to, and willing to comply with study procedures.
* Willingness to discontinue consumption of probiotic supplements and food containing added probiotics or and/or prebiotics (e.g. yoghourts, with live, active cultures or supplements).

Exclusion Criteria:

* Positive pregnancy test in women of child-bearing potential
* Pregnant or breast-feeding or planning on becoming pregnant.
* Women of child-bearing potential not using effective contraception, wich include :

Hormonal contraceptives including combined oral contraceptives, hormone birth control patch, vaginal contraceptive ring, injectable contraceptives, or hormonal implants; Intrauterine devices (IUD) or Intrauterine system (IUS); Tubal ligation; Vasectomy of partner; Double barrier method (use of physical barrier by both partners, e.g. male condom and diaphragm, male condom and cervical cap)

* Use of another investigational product within 3 months of the screening visit.
* Currently being treated for any known illnesses or conditions that may impact perceived health such as HIV/AIDS, immune modulating diseases (autoimmune, hepatitis, cancer, etc.), diabetes, kidney or liver disease, gastrointestinal diseases (e.g. gastric ulcers, Crohn's, ulcerative colitis, etc.)
* Suffered or suffering from heart attack, angina, heart arrhythmias, stroke, heart disease, thyroid problems, and diabetes requiring insulin.
* Participants with eczema, psoriasis, dermatitis or urticaria.
* Participants with soy or milk allergy.
* Participants with allergies to adhesive tape or bandages.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Evolution of the withdrawal symptoms assessed by the Mood and Physical Symptoms Scale (MPSS) | MPSS will be self-administered daily during 16 weeks
  The MPSS(M) score, corresponding to the sum of the 7 items of the MPSS mood subscale, will be compared between groups, daily between week 2 and 4 (first 2 weeks of tobacco abstinence) and week 12 and 14 (first 2 weeks after the end of NRT), and weekly for the other weeks. For weekly comparisons, an average of daily scores will be done for the respective weeks.
  The score will also be compared in time within groups, using the baseline ratings as covariates

SECONDARY OUTCOMES:
Evolution of anxiety and depression assessed by the HADS questionnaire | measured 6 times up to 16 weeks
Evolution of nicotine addiction assessed by the Fargerström Test for Nicotine Dependence | measured 3 times up to 16 weeks
Difference in tobacco abstinence between arms, determined by levels of exhaled CO and salivary cotinine dosage | measured 6 times up to 16 weeks
Evolution of body weight | measured 6 times up to 16 weeks
Evolution of food cravings | self-reported, weekly, up to 16 weeks
  Assessed by the Food Cravings Self-Questionnaire
Tolerance of the probiotics against placebo | up to 16 weeks
  Assessed by the reporting and the comparison of the Adverse events occurred in the different arms
Effect of probiotics and smoking cessation on daily bowel movement frequency and consistency, assessed by the Bristol Stool Scale | Self-reported, daily during 16 weeks
Changes in the microbiome composition of participants in the probiotic groups compared to placebo | measured 2 times up to 16 weeks
  Assessed by the analyse of the stool samples collected
Recovery of the probiotic strains in the stools | measrured 2 times up to 16 weeks
  Assessed by the change in the probiotic strains concentration in the stools samples collected in all three arms.
Evolution of nicotine addiction assessed by a visual analog scale | measured 6 times up to 16 weeks
Comparison of MPSS(Craving or C), MPSS(Physical symptoms or P), and MPSS total scores (corresponding to the sum of MPSS(M), MPSS(C) and MPSS(M) scores) | MPSS will be self-administered daily during 16 weeks
  daily comparison between week 2 and 4 (first 2 weeks of tobacco abstinence) and week 12 and 14 (first 2 weeks after the end of NRT), and weekly for the other weeks. The scores will be also compared in time within groups, using the baseline ratings as covariates. For weekly comparisons, an average of daily scores will be done for the respective weeks
Correlation between CO levels in exhaled air and salivary cotinine levels | measured 6 times up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luc Larrivée, MD, Principal Investigator — Q & T Research
Locations (1):
- Q & T Research, Sherbrooke, Quebec, Canada